CLINICAL TRIAL: NCT00487396
Title: Evaluation of Capsule Endoscopy in Patients With Suspected Crohn's Disease
Acronym: MA-51
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medtronic - MITG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: MA-51
Record Dates: First submitted 2007-06-14; First posted 2007-06-18 (Estimated); Results first posted 2012-05-16 (Estimated); Last update posted 2020-10-22 (Actual); Status verified 2020-09

CONDITIONS: Crohn's Disease
Keywords: capsule endoscopy; Crohn's disease; small bowel disease; inflammatory bowel disease; Patients with suspected small bowel Crohn's disease
MeSH Terms: conditions — Crohn Disease; Inflammatory Bowel Diseases | interventions — Capsule Endoscopy

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Capsule Endoscopy — Pillcam Platform with RAPID5 software and supporting SB2 capsules

SUMMARY:
The aim of this study is to validate the ability of Capsule Endoscopy (CE) to accurately diagnose small bowel (SB) Crohns disease in patients with symptoms of abdominal pain and diarrhea.

The primary objective of the study is to evaluate whether Capsule Endoscopy prior to colonoscopy will improve diagnosis in patients with suspected Crohns disease when compared to standard diagnostic testing.

DETAILED DESCRIPTION:
Crohn's disease is a chronic, inflammatory disorder (IBD) affecting any part of the gastrointestinal tract but frequently involves the small and large bowel. Typical presenting symptoms include abdominal pain and diarrhea. Patients with this disorder may also have extraintestinal manifestations including arthritis, uveitis and aphthous stomatitis, erythema nodosum and pyoderma gangrenosum. The etiology of Crohn's disease is unknown. It affects populations around the globe and occurs at any age but it has a predilection to affect those between the ages of 15 and 35.

While about one half of patients have involvement of the ileum and large bowel, another third have disease isolated to the small bowel. Frequently, small bowel Crohn's disease can be difficult to diagnose using the traditional methods of evaluation including colonoscopy with ileoscopy and contrast radiography. Mucosal features of Crohn's disease are often subtle and difficult to identify by small bowel follow through (SBFT). The SBFT has traditionally been relied on to evaluate the small intestine for evidence of Crohn's disease but it has been shown to have a relatively low accuracy of only 30%. This has led to delays in the diagnosis of Crohn's disease with reports ranging from one to three years.

In the past few years, capsule endoscopy has sparked renewed interest in the investigation of IBD and Crohn's disease of the small bowel. A PillCam™ SB2 capsule (Given Imaging Ltd, Yoqneam, Israel) is an ingestible, disposable video camera that transmits high quality images of the small intestinal mucosa. This enables the small intestine to be readily accessible to physicians investigating for the presence of small bowel disorders which in the past was inaccessible to physicians. A number of small pilot studies demonstrated capsule endoscopy efficacy in diagnosing SB Crohn's disease. Diagnostic yields of 70% have been reported in small series of studies performed in suspected small bowel Crohn's disease.

This study is designed to determine the yield and clinical impact of Capsule Endoscopy (CE) in detecting suspected IBD and suspected Crohn's Disease of the small bowel when compared to SBFT.

ELIGIBILITY:
Inclusion Criteria:

* Patients ages 10-65 years, inclusive

  * Patient suffers from either

    * diarrhea for more than 6 weeks and less than 3 years and/or
    * abdominal pain for more than 6 weeks and less than 3 years and/or
    * extra-luminal manifestations of IBD including: erythema nodosum, pyoderma gangrenosum, arthritis, peri-anal disease, uveitis, aphthous stomatitis
  * Patient suffers from at least one of the symptoms / lab abnormalities listed below:

    * Positive inflammatory marker (ESR, CRP, thrombocytosis, leukocytosis, fecal lactoferrin, fecal alpha-1 antitrypsin) within 3 months prior to enrollment
    * Unexplained anemia (less than normal limits) within 3 months prior to enrollment
    * Hypoalbuminemia (<3.5 g/dl) within 3 months of enrollment
    * Positive ASCA within 3 months of enrollment
    * Abnormal white blood cell scan with in 3 months of enrollment
    * Stool negative for O&P (C&S) within 3 months of enrollment
    * Recurrent Fevers
    * Unexplained weight loss, failure to thrive in children
    * Gastro-intestinal bleeding including melena and/or hematochezia and/or FOBT positive.
    * Chronic perianal disease (fistula, fissure, peri-rectal abscess)
    * Abnormal small bowel SBFT and/or enteroclysis and/or abdominal CT not conclusively diagnostic for IBD
  * Patient is indicated for Ileo-Colonoscopy
  * Patient or legal guardian agrees to sign consent form

Exclusion criteria:

* Indeterminate Colitis where the purpose is only to make a definitive diagnosis and where the inclusion criteria are not otherwise met
* Known intestinal obstruction or current obstructive symptoms, such as severe abdominal pain with accompanying nausea or vomiting.
* Definite long stricture seen on radiological exam.
* Suspected GI stricture, followed by agile™ study that could not prove patency of the GI tract.
* Known history of small bowel Crohn's Disease
* Current treatment for active IBD
* Positive Anti-tTG or anti-endomysial antibody
* Any of the following work-up within 1 year of study entry: Capsule Endoscopy, Colonoscopy and Upper GI/SBFT.
* Non-steroidal anti-inflammatory drugs including Aspirin, (twice weekly or more) during the 4 weeks preceding enrollment
* Patient is pregnant

Ages: 10 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2007-09; Primary Completion 2010-10 (Actual); Study Completion 2010-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Leighton, MD, Principal Investigator — Mayo Clinic; Peter Legnani, MD, Principal Investigator — Private Practice New York, New York
Locations (11):
- United States (8):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - Atlanta Gastroenterology, Atlanta, Georgia
  - Stan Cohen, Atlanta, Georgia
  - John Hopkins - Department of Medicine, Baltimore, Maryland
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - Minnesota Gastroenterology Associates, Plymouth, Minnesota
  - Private Practice, New York, New York
  - Thomas Jefferson University, Philadelphia, Pennsylvania
- McGill University Health Center, Montreal, Quebec, Canada
- Rambam Medical Center, Haifa, Israel
- Malmo University Hospital UMAS, Malmo, Sweden

REFERENCES:
- [Derived] Leighton JA, Gralnek IM, Cohen SA, Toth E, Cave DR, Wolf DC, Mullin GE, Ketover SR, Legnani PE, Seidman EG, Crowell MD, Bergwerk AJ, Peled R, Eliakim R. Capsule endoscopy is superior to small-bowel follow-through and equivalent to ileocolonoscopy in suspected Crohn's disease. Clin Gastroenterol Hepatol. 2014 Apr;12(4):609-15. doi: 10.1016/j.cgh.2013.09.028. Epub 2013 Sep 27. PMID 24075891

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study started on September 2007 and data collection completed on October 2010. Study conducted in 10 clinical sites (hospitals and private clinics) in the USA, Sweden, Canada and Israel
Pre-assignment Details: 98 patients enrolled in this study. 18 cases excluded due to the following: 15 cases were excluded due to noncompliance with the protocol.
  1 patient withdrew consent before any study procedure.
  1 patient could not ingest the capsule.
  1 patient refused to undergo the ileocolonoscopy and SBFT. Therefore 80 patients were included in the analysis
Groups:
- SB Capsule Then Standard Ileocolonoscopy: Capsule endoscopy was ingested .The purpose was to detect patients with crohn Patients subsequently had standard ileocolonoscopy and small bowel follow through as comparison.
Period: Overall Study
Arm/Group | SB Capsule Then Standard Ileocolonoscopy
Started | 98
Completed | 95
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: 98 patients enrolled in this study. 18 cases excluded due to the following: 15 cases were excluded due to noncompliance with the protocol.
  1 patient withdrew consent before any study procedure.
  1 patient could not ingest the capsule.
  1 patient refused to undergo the ileocolonoscopy and SBFT. Therefore 80 patients were included in the analysis
Groups:
- SB Capsule Then Standard Ileocolonoscopy: Capsule endoscopy was ingested.The purpose was to detect patients with Crohn's Disease. Patients subsequently had standard ileocolonoscopy and small bowel follow through as comparison.
Arm/Group | SB Capsule Then Standard Ileocolonoscopy
Number analyzed (Participants) | 80
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 20
  Between 18 and 65 years | 60
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.35 (13.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38
  Male | 42
Region of Enrollment [Number; unit: participants]
  United States | 46
  Israel | 20
  Sweden | 14

OUTCOME MEASURES:

1. Primary Outcome: Diagnostic Yield in Suspected Crohn's Patients (CE Prior to IC vs. IC and SBFT)
Description: To evaluate whether capsule endoscopy (CE) prior to ileocolonoscopy (IC) improves the diagnostic yield in patients with suspected Crohn's disease when compared to IC and SBFT. McNemar test was preformed in order to evaluate the diagnostic yield of IC combined with CE as compared to the diagnostic yield of IC combined with SBFT.
Time Frame: four months from enrollment
Population: The number of found and missed pathologies (i.e. ulcers, lesions, etc.) were calculated for the combination of procedures.
Measure: Number; unit: percentage of yield
Units Other Than Participants: pathologies
Groups:
- PillCam SB Followed by Ileo Colonoscopy: Ingestible capsule equipped with an endoscope with one imagers, before ileo-colonoscopy.
- Small Bowel Follow Through (SBFT) and Ileo-colonoscopy: Following ingestible capsule, same patients also underwent ileo-colonoscopy (IC) and small bowel follow through (SBFT).
Arm/Group | PillCam SB Followed by Ileo Colonoscopy | Small Bowel Follow Through (SBFT) and Ileo-colonoscopy
Number analyzed (Participants) | 74 | 74
Number analyzed (pathologies) | 110 | 110
percentage of yield | 97.3 | 57.3
Statistical Analysis 1: Comparison: PillCam SB Followed by Ileo Colonoscopy vs Small Bowel Follow Through (SBFT) and Ileo-colonoscopy; Pathologies were including in the analysis as follows: * combination of CE+IC procedures but not detected by the combination of SBFT+IC procedures were marked as "CE+IC new finding" ; * Pathologies detected by the combination of SBFT+IC procedures but not detected by the combination of CE+IC procedures were marked as "SBFT+IC new finding" event; * Pathologies detected by the combination of CE+IC procedures and by the combination of SBFT+IC procedures were marked as "same findings" event; Test type: Other; p < 0.0001, McNemar

2. Secondary Outcome: Diagnostic Yield (CE vs. SBFT)
Description: McNemar test was preformed in order to evaluate the diagnostic yield of PillCam SB (CE) as compared to the diagnostic yield of small bowel follow through (SBFT).
Time Frame: four months from enrollment
Population: as for outcome 1
Measure: Number; unit: percentage of yield
Units Other Than Participants: pathologies
Groups:
- Pill Cam SB Capsule (CE); Small Bowel Follow Through (SBFT): Capsule endoscopy was ingested. The purpose was to detect patients with crohn's disease. Patients subsequently had standard ileocolonoscopy and small bowel follow through as comparison.
Arm/Group | Pill Cam SB Capsule (CE) | Small Bowel Follow Through (SBFT)
Number analyzed (Participants) | 72 | 72
Number analyzed (pathologies) | 43 | 43
percentage of yield | 93.0 | 25.6
Statistical Analysis 1: Comparison: Pill Cam SB Capsule (CE) vs Small Bowel Follow Through (SBFT); For each category, the numbers of found and missed pathologies were including in the analysis as follows: * Pathologies detected by CE procedure but not detected by SBFT procedure were marked as "CE new finding" event; * Pathologies detected by SBFT procedure but not detected by CE procedure were marked as "SBFT new finding" event; * Pathologies detected by both procedures (i.e., CE and SBFT) were marked as "same findings" event; Test type: Other; p < 0.0001, McNemar

3. Secondary Outcome: Diagnostic Yield (CE vs. IC)
Description: McNemar test was preformed in order to evaluate the diagnostic yield of PillCam SB (CE) as compared to the diagnostic yield of ileocolonoscopy (IC).
Time Frame: four months from enrollment
Population: as for outcome 1
Measure: Number; unit: percentage of yield
Units Other Than Participants: pathologies
Groups:
- PillCam SB Capsule; Standard Ileocolonoscopy (IC): Capsule endoscopy was ingested.The purpose was to detect patients with crohn's disease. Patients subsequently had standard ileocolonoscopy and small bowel follow through as comparison.
Arm/Group | PillCam SB Capsule | Standard Ileocolonoscopy (IC)
Number analyzed (Participants) | 80 | 80
Number analyzed (pathologies) | 61 | 61
percentage of yield | 49.2 | 70.5
Statistical Analysis 1: Comparison: PillCam SB Capsule vs Standard Ileocolonoscopy (IC); Pathologies were including in the analysis as follows: * Pathologies detected by CE procedure but not detected by IC procedure were marked as "CE new finding" event; * Pathologies detected by IC procedure but not detected by CE procedure were marked as "IC new finding" event; * Pathologies detected by both procedures (i.e., CE and IC) were marked as "same findings" event; Test type: Other; p = 0.085, McNemar

ADVERSE EVENTS:
Time Frame: Adverse event monitoring was performed for each visit during the visit and the following 1-3 days. Participation lasted for up to 12 months.
Groups:
- Adverse Events: All subjects received both the capsule endoscopy procedure and the ileocolonoscopy procedure
Arm/Group | Adverse Events
All-Cause Mortality (participants affected / at risk) | 0/80
Serious Adverse Events (participants affected / at risk) | 1/80
Other Adverse Events (participants affected / at risk) | 8/80
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adverse Events (N=80)
Capsule Retention (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adverse Events (N=80)
Weakness (General disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 1 (1)
Capsule retention (Product Issues) | 2 (2)
Blood in stool (Gastrointestinal disorders) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1)
dehydration (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No